CLINICAL TRIAL: NCT05883917
Title: Clinical Utility of Robot-Assisted Gait Training in Patients With Spinal Cord Injury Caused by Electrical Burns: A Case Report
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Hangang Sacred Heart Hospital, Hangang Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-15
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Gait Disorder, Sensorimotor; Burns; Spinal Cord Injuries
MeSH Terms: conditions — Gait Disorders, Neurologic; Burns; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Gait training using SUBAR® (Cretem, Korea) proceeded by adjusting parameters (gait speed, step length, and degree of knee flexion) according to the patient's leg length and gait function. The parameters were set to the maximum levels tolerated by the patient. The patients underwent 30 min of robot-assisted training using SUBAR® with 30 min of conventional physiotherapy, 5 days a week for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- robot assisted gait training (Experimental): Gait training using SUBAR® (Cretem, Korea) proceeded by adjusting parameters (gait speed, step length, and degree of knee flexion) according to the patient's leg length and gait function. The parameters were set to the maximum levels tolerated by the patient. The patients underwent 30 min of robot-assisted training using SUBAR® with 30 min of conventional physiotherapy, 5 days a week for 12 weeks.
  Interventions: Procedure: robot assisted gait training

INTERVENTIONS:
Procedure: robot assisted gait training — Gait training using SUBAR® (Cretem, Korea) proceeded by adjusting parameters (gait speed, step length, and degree of knee flexion) according to the patient's leg length and gait function. The parameters were set to the maximum levels tolerated by the patient. The patients underwent 30 min of robot-assisted training using SUBAR® with 30 min of conventional physiotherapy, 5 days a week for 12 weeks.

SUMMARY:
Robot-assisted gait training has been effective in several diseases. Nevertheless, evidence supporting the efficacy of such training in burn patients remains insufficient. This report aimed to evaluate the effect of robot-assisted gait training in burn patients with spinal cord injuries caused by electrical trauma.

We will report a case of two patients who underwent 30 min of robot-assisted gait training using SUBAR® (Cretem, Korea) with 30 min of conventional physiotherapy, 5 days a week for 12 weeks.

DETAILED DESCRIPTION:
Robot-assisted gait training has been effective in several diseases. Nevertheless, evidence supporting the efficacy of such training in burn patients remains insufficient. This report aimed to evaluate the effect of robot-assisted gait training in burn patients with spinal cord injuries caused by electrical trauma.

Gait training using SUBAR® (Cretem, Korea) proceeded by adjusting parameters (gait speed, step length, and degree of knee flexion) according to the patient's leg length and gait function. The parameters were set to the maximum levels tolerated by the patient. The patients underwent 30 min of robot-assisted training using SUBAR® with 30 min of conventional physiotherapy, 5 days a week for 12 weeks.

All measurements were assessed before training (0 week) and after training (12 weeks). The American Spinal Injury Association (ASIA) lower extremity motor subscale score (LEMS; range 0-50) was used to evaluate motor function. LEMS is the sum of bilateral lower extremity key muscle power, ranging from total paralysis (0) to normal active movement with a full range of motion against gravity and maximum resistance (5), with a total possible score of 50. The passive range of motions (ROMs) of different joints (hip, knee, and ankle) were measured using a goniometer. The ambulatory motor index (AMI; range 0-30), which predicts ambulatory capability, was measured by evaluating muscles of hip flexion, hip abduction, hip extension, knee extension, and knee flexion on both sides. Functional Ambulation Categories (FAC) scores and 6-min walking test (6MWT) distances were measured to evaluate functional recovery. FAC was evaluated based on a 6-point scale, from 0 (the patient cannot walk or can only walk with the assistance of two people) to 5 (the patient can walk independently). 6MWT followed the standardised guidelines, and the walking course was 20 m. The patients were instructed to walk as far as possible in 6 min .

ELIGIBILITY:
Inclusion Criteria:

* electrical burn
* spinal cord injury
* aged > 18 years
* aged <75 years
* ≤ 1 functional ambulation category (FAC) score of ≤3

Exclusion Criteria:

* had fourth-degree burns (involving muscles, tendons, and bone injuries)
* had musculoskeletal diseases (fracture, amputation, rheumatoid arthritis, and degenerative joint diseases) involving the burned lower extremity.
* cognitive disorders
* intellectual impairment before burn injury
* serious cardiac dysfunction
* skin disorders that could be worsened by RAGT
* severe pain who were unable to undergo rehabilitation programs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association | 12 weeks

SECONDARY OUTCOMES:
lower extremity motor subscale score (LEMS; range 0-50) | 12 weeks
  LEMS is the sum of bilateral lower extremity key muscle power, ranging from total paralysis (0) to normal active movement with a full range of motion against gravity and maximum resistance (5), with a total possible score of 50
passive range of motions | 12 weeks
  The passive range of motions (ROMs) of different joints (hip, knee, and ankle) were measured using a goniometer
The ambulatory motor index (AMI; range 0-30) | 12 weeks
  predicts ambulatory capability, was measured by evaluating muscles of hip flexion, hip abduction, hip extension, knee extension, and knee flexion on both sides

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ohn SH, Kim DY, Shin JC, Kim SM, Yoo WK, Lee SK, Park CH, Jung KI, Jang KU, Seo CH, Koh SH, Jung B. Analysis of high-voltage electrical spinal cord injury using diffusion tensor imaging. J Neurol. 2013 Nov;260(11):2876-83. doi: 10.1007/s00415-013-7081-1. Epub 2013 Sep 4. PMID 24002417
- [Result] Cheung EYY, Ng TKW, Yu KKK, Kwan RLC, Cheing GLY. Robot-Assisted Training for People With Spinal Cord Injury: A Meta-Analysis. Arch Phys Med Rehabil. 2017 Nov;98(11):2320-2331.e12. doi: 10.1016/j.apmr.2017.05.015. Epub 2017 Jun 20. PMID 28645768
- [Derived] Lee SY, Seo CH, Ch YS, Kim Y, Yoon Y, Joo SY. Exoskeleton Robot Training in Two Patients with an Electrical Burn and Septic Arthritis: A Case Report. J Burn Care Res. 2025 Aug 12;46(3):646-651. doi: 10.1093/jbcr/irae205. PMID 39851068